CLINICAL TRIAL: NCT05681494
Title: Assessment of Postoperative Pain and Treatment Success After Vital Pulp Therapy Versus Root Canal Treatment in Mature Permanent Mandibular Molars With Irreversible Pulpitis: A Randomized Controlled Trial
Brief Title: Assessment of Pain and Treatment Success After VPT Versus RCT in Mature Permanent Mandibular Molars With SIP: A RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amany Ibrahiem Ahmed Mohamed, Ph.D. degree candidate, Department of Endodontics, Faculty of Dentistry, Cairo university., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 28/12/2022
Record Dates: First submitted 2022-12-28; First posted 2023-01-12 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Symptomatic Irreversible Pulpitis
Keywords: SIP
MeSH Terms: interventions — Pulpotomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Root canal treatment (Active Comparator): after access cavity preparation, the working length will be determined. chemo-mechanical preparation will be done, and teeth will be obturated. final restoration will be placed.
  Interventions: Procedure: Root canal treatment
- Vital pulp therapy (Experimental): exposed pulp will be capped with 3 mm calcium silicate material
  Interventions: Procedure: Vital pulp therapy

INTERVENTIONS:
Procedure: Root canal treatment — after access cavity preparation, the working length will be determined. chemo-mechanical preparation will be done, and teeth will be obturated. final restoration will be placed.
  Other Names: RCT, Full pulpectomy
  Arms: Root canal treatment
Procedure: Vital pulp therapy — exposed pulp will be capped with 3 mm calcium silicate material
  Other Names: pulpotomy
  Arms: Vital pulp therapy

SUMMARY:
Assessment of postoperative pain and treatment success after vital pulp therapy versus root canal treatment in mandibular molar with signs and symptoms of irreversible pulpitis. the null hypothesis, there is no difference will be observed in the pain level and treatment success between two treatments.

DETAILED DESCRIPTION:
After proper clinical and radiographic examination. Teeth will be anesthetized and isolated using a rubber dam. The operative field will be disinfected. Total caries removal will be done from outside making margin caries free to inside. the new diamond bur will be used to remove the last layer and exposed the pulp tissue. Exposed pulp will be inspected under a dental operating microscope and hemostasis will be obtained. The teeth will be randomized into 2 intervention groups (VPT or RCT). Treatment will be finalized, and teeth will be restored with resin-modified glass ionomer followed by composite resin at the same appointment. Ibuprofen 400mg will be prescribed to the patient if needed. Patients will be asked to record postoperative pain after treatment on the pain score sheet.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients.
* Patient's age range more than 15 years.
* Mature permanent mandibular molars with deep caries.
* Clinical diagnosis of symptomatic irreversible pulpitis.
* Teeth with no need for the post.
* Healthy periodontium and mobility within normal limits.
* Patients who can understand the pain scale and can sign the informed consent

Exclusion Criteria:

* Teeth with a negative response to vitality testing.
* Teeth with furcal bone loss.
* Teeth with sinus tract
* Teeth with swelling.
* Teeth with a non-restorable crown.
* Teeth with immature roots.
* Teeth with no pulp exposure even after caries excavation.
* History of analgesic intake in the previous week.
* History of antibiotic intake in the previous month.
* Insufficient bleeding after pulp exposure suggestive of partial necrosis of the pulp.
* Inability to control bleeding within 10 min.
* Radiographic evidence of external or internal root resorption vertical root fracture, perforation, calcification.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-02-26 (Estimated); Primary Completion 2023-07-26 (Estimated); Study Completion 2024-06-26 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | at 6 hours postoperative
  postoperative pain will be recorded by patient using NRS

SECONDARY OUTCOMES:
Intensity of postoperative pain | at 24, 48 hours and 7 days
  postoperative pain will be recorded by patient using NRS
Treatment success | at 3,6,12 months
  clinical and radiographic success

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed S Elsheshtawy, Study Director — Lecturer, Department of Endodontics, Faculty of Dentistry, Cairo university.

REFERENCES:
- [Background] Taha NA, Al-Rawash MH, Imran ZA. Outcome of full pulpotomy in mature permanent molars using 3 calcium silicate-based materials: A parallel, double blind, randomized controlled trial. Int Endod J. 2022 May;55(5):416-429. doi: 10.1111/iej.13707. Epub 2022 Mar 17. PMID 35152464
- [Background] Santos JM, Pereira JF, Marques A, Sequeira DB, Friedman S. Vital Pulp Therapy in Permanent Mature Posterior Teeth with Symptomatic Irreversible Pulpitis: A Systematic Review of Treatment Outcomes. Medicina (Kaunas). 2021 Jun 3;57(6):573. doi: 10.3390/medicina57060573. PMID 34205149
- [Background] Taha NA, Al-Khatib H. 4-Year Follow-up of Full Pulpotomy in Symptomatic Mature Permanent Teeth with Carious Pulp Exposure Using a Stainproof Calcium Silicate-based Material. J Endod. 2022 Jan;48(1):87-95. doi: 10.1016/j.joen.2021.09.008. Epub 2021 Sep 24. PMID 34563506
- [Background] Asgary S, Eghbal MJ, Shahravan A, Saberi E, Baghban AA, Parhizkar A. Outcomes of root canal therapy or full pulpotomy using two endodontic biomaterials in mature permanent teeth: a randomized controlled trial. Clin Oral Investig. 2022 Mar;26(3):3287-3297. doi: 10.1007/s00784-021-04310-y. Epub 2021 Dec 2. PMID 34854987